CLINICAL TRIAL: NCT00485199
Title: Pneumatic Retinopexy Versus Vitrectomy With Gas for Retinal Detachment Due to Myopic Macular Hole
Acronym: RDMH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RDMH2007-china
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Last update posted 2007-06-12 (Estimated); Status verified 2007-06

CONDITIONS: Retinal Detachment
Keywords: Pneumatic Retinopexy; vitrectomy; retinal detachment; macular hole; treatment; multi-center; Retinal Detachment due to Myopic Macular hole
MeSH Terms: conditions — Retinal Detachment; Retinal Perforations | interventions — Vitrectomy; Gases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Pneumatic Retinopexy
Procedure: Vitrectomy with Gas

SUMMARY:
To undertake a prospective randomized clinical study for treating retinal detachment due to myopic macular holes, utilizing pneumatic retinopexy versus pars plana vitrectomy with gas tamponade.To determine the efficiency of pneumatic retinopexy with C3F8 in the treatment of retinal detachment due to myopic macular hole.

DETAILED DESCRIPTION:
Retinal detachment caused by macular hole predominantly happened in high myopic eyes. This is a common type of retinal detachment in Asia and often seen in the old people aged around 50 ~ 60, mainly in female. Treatment of retinal detachment due to macular holes has changed over the years, and several methods have been described. Some surgeons have used transscleral diathermy or cryotherapy or laser photocoagulation and drainage subretinal fluid without sclera buckling, other surgeons have used radial silicone explants beneath the macular combined with cryo, diathermy or laser. This method entails the difficulty of placing sclera sutures far posterior, especially hazardous if there is a posterior staphyloma with very thin sclera. Besides the technically difficult, the extensive macular scarring caused by different coagulations limited the functional result to peripheral vision only. Because of this, it is not generally used in the initial treatment.

In 1982, Gonvers and Machemer4 proposed a new treatment technique that combined pars plana vitrectomy (PPV), partial air-fluid exchange, and face down positioning for 24 hours. Since then vitrectomy with gas tamponade become the most common procedure for retinal detachment with macular hole.

In 1984, Miyake performed a simple gas injection into the vitreous followed by a face-down position. The effective of this simplified method was then reported by many observers.But these studies may have insufficiency because of small sample, nonrandomized, no defined eligibility criteria for patients selection.

Intraocular gas tamponade with or without pars plana vitrectomy (PPV) has commonly been performed nowadays. We conducted a multicenter randomized controlled clinical trial to compare their anatomic results and visual outcomes of both surgical techniques, to estimate the efficiency of both surgical methods in the treatment of retinal detachment with myopic macular hole.

ELIGIBILITY:
Inclusion Criteria:

* retinal detachment due to myopic macular hole.
* The ability to give informed consent and to return for follow-up visit for 12 months

Exclusion Criteria:

* retinal detachment with macular hole and peripheral hole/tear
* retinal detachment with severe proliferative vitreoretinopathy
* retinal detachment with choroidal detachment or rupture
* traction retinal detachment due to retinal vascular disease
* had vitrectomy in the past
* macular hole without retinal detachment
* foveal schiesis without retinal detachment
* secondary macular hole with retinal detachment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2005-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
BCVA improvement,anatomic success | 1,3,6,9, and 12 months after treatment

SECONDARY OUTCOMES:
costs of treatment | right after the treatment
complication | 1,3,6,9, 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxin Li, professor, Study Chair — Peking University; Jialiang Zhao, professor, Principal Investigator — Eye Institute of Peking Union Hospital, Peking Union Medical College; Wenji Wang, professor, Principal Investigator — Department of ophthalmology of Eye Ear Nose Throat Hospital, Fudan University, Shanghai; Shibo Tang, professor, Principal Investigator — Zhong Shan Ophthalmic Center, Sun Yat-sen University
Locations (14):
- China (14):
  - Department of ophthalmology of People Hospital, Peking University, Beijing, Beijing Municipality
  - Department of ophthalmology of Beijing Hospital, Beijing, Beijing Municipality
  - Department of ophthalmology of Beijing Tong Ren Hospital, Beijing, Beijing Municipality
  - Department of ophthalmology of China PLA General Hospital, Beijing, Beijing Municipality
  - Peking Eye Center of the third affiliated Hospital of Peking University, Beijing, Beijing Municipality
  - Zhong Shan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong
  - Department of ophthalmology of The Second affiliated Xiang Ya Hospital, Central South University, Changsha, Hunan
  - Department of ophthalmology of The First affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Department of ophthalmology of The First affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Eye Institute, Qingdao, Shandong
  - Department of ophthalmology of EENT Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Department of ophthalmology of The First affiliated People Hospital of Shang Hai Jiao Tong University, Shanghai, Shanghai Municipality
  - Department of ophthalmology of West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Eye Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Schwartz SG, Flynn HW Jr, Wang X, Kuriyan AE, Abariga SA, Lee WH. Tamponade in surgery for retinal detachment associated with proliferative vitreoretinopathy. Cochrane Database Syst Rev. 2020 May 13;5(5):CD006126. doi: 10.1002/14651858.CD006126.pub4. PMID 32408387